CLINICAL TRIAL: NCT06056388
Title: Is the Accuracy of Immediate Implant Placement Using Dynamic Navigation Affected by Fixture Thread Depth?: A Randomized Controlled Trial
Brief Title: Effect of Fixture Thread Depth on Accuracy of Immediate Implant Placement Using Dynamic Navigation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDC-23-1
Record Dates: First submitted 2023-09-03; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-08

CONDITIONS: Tooth Loss; Partial-edentulism
Keywords: Computer-Assisted Surgery; Dental Implants
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Deep-threaded implants (Active Comparator): Straumann BLX implants
  Interventions: Device: Straumann BLX implant
- Regular-threaded implants (Placebo Comparator): Straumann BLT implants
  Interventions: Device: Straumann BLT implant

INTERVENTIONS:
Device: Straumann BLX implant — Implant system with a deep fixture thread depth.
  Arms: Deep-threaded implants
Device: Straumann BLT implant — Implant system with a regular fixture thread depth.
  Arms: Regular-threaded implants

SUMMARY:
The goal of this clinical trial is to compare the placement accuracy in immediately placed implants using dynamic navigation between deep-threaded and regular-threaded implants in partially edentulous patients. The main question it aims to answer is: is there a difference in implant placement accuracy between deep-threaded and regular-threaded implants using dynamic navigation? Participants will receive implants placed immediately under dynamic guidance. Researchers will compare type of implant thread (Straumann BLT versus Straumann BLX) to see if there are significant differences in placement accuracy.

DETAILED DESCRIPTION:
The initial visit will comprise a thorough clinical examination and panoramic radiograph acquisition. Hopeless teeth resulting from trauma, periapical abscess, and periodontitis will be evaluated to see if extraction indications are met. When extraction indications were met, patients will be evaluated for suitable bone height for immediate implant placement. When bone height was suitable, patients will be asked to take a preoperative CBCT scan.

After tooth condition and bone volume evaluations, patients with adequate bone volume for immediate implant placement will be enrolled and randomly assigned to one of two groups: deep-threaded or regular-threaded.

The following implant placement accuracy parameters will be recorded using postoperative intraoral scanning superimposition: Global platform deviation (measured in millimeters), lateral platform deviation (measured in millimeters), global apex deviation (measured in millimeters), apex depth deviations (measured in millimeters), and angular deviation (measured in degrees). Primary implant stability will be measured immediately after implant insertion and measured in both insertion torque value and implant stability quotient. Radiographic bone-implant contact will be measured with a 3D implant model reconstruction method using coDiagnostiX and the contact area will be calculated using 3-matic Research as previously reported. Marginal bone loss will be measured using ImageJ with periapical radiographs taken 3 months and 1-year post-op. Implant survival will be monitored starting from the final prosthesis delivery onwards. Complications (biological, technical, and implant loss) will be recorded accordingly. Patient satisfaction will be documented with a Mandarin Chinese version of the Short Form Patient Satisfaction Questionnaire (PSQ-18) upon final prosthesis delivery.

ELIGIBILITY:
Inclusion Criteria:

* Hopeless teeth that require extraction
* No systemic diseases
* Smoking (<10 cigarettes/day)
* Full-mouth bleeding and full-mouth plaque index lower than or equal to 25%
* Fresh extraction sockets with at least 3 fully intact socket walls
* At least 4 mm of bone beyond the root apex
* Meets one of the following:
* Single immediate placement site in the maxillary esthetic zone [15-25 (FDI classification)].
* Two or more nonconsecutive immediate placement sites in the maxillary esthetic zone [15-25 (FDI classification)].
* Two or more consecutive immediate placement sites in the maxillary esthetic zone [15-25 (FDI classification)].

Exclusion Criteria:

* General medical (American Society of Anesthesiologists, ASA, class III or IV) and/or psychiatric contraindications
* Pregnancy or nursing
* Any interfering medication such as steroid therapy or bisphosphonate therapy
* Alcohol or drug abuse
* Heavy smoking (>10 cigarettes/day)
* Radiation therapy to head or neck region within 5 years
* Untreated periodontitis
* Refuse to participate in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-31 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Placement accuracy measured as global platform deviation in millimeters and assessed by DCarer or coDiagnostiX | Postoperative (Day 1-5)
  Sufficiently described in the Title
Placement accuracy measured as lateral platform deviation in millimeters and assessed by DCarer or coDiagnostiX | Postoperative (Day 1-5)
  Sufficiently described in the Title
Placement accuracy measured as global apex deviation in millimeters and assessed by DCarer or coDiagnostiX | Postoperative (Day 1-5)
  Sufficiently described in the Title
Placement accuracy measured as apex depth deviations in millimeters and assessed by DCarer or coDiagnostiX | Postoperative (Day 1-5)
  Sufficiently described in the Title
Placement accuracy measured as angular deviation in degrees and assessed by DCarer or coDiagnostiX | Postoperative (Day 1-5)
  Sufficiently described in the Title

SECONDARY OUTCOMES:
Level of primary implant stability measured in insertion torque (ITV) using a Torq Control | Intraoperative (Day 0)
  Sufficiently described in the Title
Level of primary implant stability measured in implant stability quotient (ISQ) using an Osstell Beacon | Intraoperative (Day 0)
  Sufficiently described in the Title
Amount of radiographic bone-implant contact measured in millimeters using 3-matic Research | Postoperative (Day 1-5)
  Sufficiently described in the Title
Amount of marginal bone loss measured in millimeters using periapical radiographs | Postoperative (1 year)
  Sufficiently described in the Title
Rate of implant survival measured in percentage | Postoperative (4 months & 1 year)
  Sufficiently described in the Title
Number of participants with biological or technical complications | Postoperative (Up to 1 year)
  Sufficiently described in the Title
Level of patient satisfaction measured using the Short Form Patient Satisfaction Questionnaire | Postoperative (4 months & 1 year)
  Minimum value: 18; Maximum value: 90; Higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Yiqun Wu, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University

REFERENCES:
- [Result] Skjerven H, Olsen-Bergem H, Ronold HJ, Riis UH, Ellingsen JE. Comparison of postoperative intraoral scan versus cone beam computerised tomography to measure accuracy of guided implant placement-A prospective clinical study. Clin Oral Implants Res. 2019 Jun;30(6):531-541. doi: 10.1111/clr.13438. Epub 2019 May 12. PMID 31002415
- [Result] Gu Y, Zhang D, Tao B, Wang F, Chen X, Wu Y. A novel technique to quantify bone-to-implant contact of zygomatic implants: a radiographic analysis based on three-dimensional image registration and segmentation. Dentomaxillofac Radiol. 2023 Jan;52(2):20220210. doi: 10.1259/dmfr.20220210. Epub 2023 Jan 16. PMID 36645052